CLINICAL TRIAL: NCT05437380
Title: The Value of Peritumoral Microbubbles and Contrast-enhanced Ultrasonography to Detect and Biopsy Sentinel Lymph Nodes in Head and Neck Squamous Cell Carcinoma
Brief Title: Peritumoral Microbubbles and CEUS for SLN Detection and Biopsy in HNSCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSKY-2022-019-02
Record Dates: First submitted 2022-06-26; First posted 2022-06-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-05

CONDITIONS: Sentinel Lymph Node; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEUS (Experimental)
  Interventions: Diagnostic Test: peritumoral microbubbles and contrast-enhanced ultrasonography

INTERVENTIONS:
Diagnostic Test: peritumoral microbubbles and contrast-enhanced ultrasonography — Inject 1ml microbubbles around the tumors. Then detect lymph vessel and lymph nodes under contrast-enhanced ultrasonography.

SUMMARY:
Head and neck squamous cell carcinoma is the sixth most common malignant tumor in the world. Cervical lymph node metastasis is frequently encounted on the date of diagnosis. Surgical resection is one of the most important treatment methods for head and neck squamous cell carcinoma with or without lymph node metastasis. At present, for cN0 patients, prophylactic neck dissection is recommended for squamous cell carcinoma originating in suprglottic, hypopharyngeal and oropharyngeal areas et al. Related studies reported that less than 30% of patients with cN0 were confirmed to have lymph node metastasis in postoperative pathological examination, who underwent neck dissection. Unnecessary neck dissection may increase complication incidence, such as neurovascular injury, chylous leakage, sialosyrinx. Accurate preoperative assessment is helpful to reduce unnecessary neck dissection. Sentinel lymph node biopsy were proved to be effective in reducing prophylactic lymph node dissection in breast cancer, melanoma and other malignant tumors. Compared with γ probe detection and indolyanine green injection, microbubble and contrast-enhanced ultrasound has no radiation and disturbance to resection margins in sentinel lymph nodes detection. Furthermore, surgeons could conduct lymph node puncture biopsy simultaneously under ultrasound guidance, which can further minimize surgical trauma. At present, the role of microbubble and contrast-enhanced ultrasound in sentinel lymph node detection and biopsy is rarely reported in head and neck squamous cell carcinoma. This study aims to explore the accuracy of peritumoral microbubbles and contrast-enhanced ultrasound for sentinel lymph nodes biopsy in predicting cervical lymph node metastasis in head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70;
* Pathological biopsy indicated head and neck squamous cell carcinoma;
* MR/CT examination indicate no suspected cervical lymph node metastasis;
* The patient intent to perform primary focal resection and unilateral/bilateral neck dissection at our center;
* agree to participate in clinical trials and sign informed consent.

Exclusion Criteria:

* allergic to microbubbles contrast agents;
* patients who cannot tolerate surgery;
* enlarged cervical lymph node in palpation or suspected cervical lymph node metastasis indicated in MR/CT examination;
* distant metastasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 4 years
  diagnostic accuracy=(true positive+true negative)/(true positive+true negative+false positive+false negative)

CONTACTS AND LOCATIONS:
Overall Officials: Huang Xiaoming, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China